CLINICAL TRIAL: NCT04958811
Title: A Phase II Open-label Multi-cohort Study Evaluating the Efficacy of Tiragolumab With Atezolizumab Plus Bevacizumab in Previously-Treated Advanced Non-squamous NSCLC
Brief Title: Tiragolumab With Atezolizumab Plus Bevacizumab in Previously-Treated Advanced Non-squamous NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003943
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Non-squamous Non-small-cell Lung Cancer
Keywords: Lung Cancer; Non-squamous Non-small-cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Tiragolumab; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tiragolumab plus atezolizumab and bevacizumab (Experimental): Tiragolumab 600mg IV will be administered together with atezolizumab 1200mg IV and bevacizumab 15mg/kg IV every 3 weeks (q3w) until progressive disease or unacceptable toxicity.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Tiragolumab — 600mg IV administered every 3 weeks.
Drug: Atezolizumab — 1200mg IV administered every 3 weeks.
Drug: Bevacizumab — 15mg/kg IV administered every 3 weeks.

SUMMARY:
To evaluate the efficacy of tiragolumab with atezolizumab and bevacizumab in previously-treated advanced non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF)
* Age ≥ 18 years at time of signing ICF
* Ability to comply with the study protocol, in the investigator's judgment
* Histologically or cytologically confirmed advanced non-squamous NSCLC that is not amenable to definitive therapy
* Tumor PD-L1 expression (TPS ≥ 1%) (cohort A only)
* EGFR, ALK, ROS1 wild-type (cohort A only)
* Confirmed activating alteration in EGFR (cohort B only)
* Disease progression during or following treatment with anti-PD(L)1 containing therapy (cohort A only)
* Disease progression during or following treatment with appropriate EGFR targeted therapy (cohort B only)
* Measurable disease per RECIST v1.1
* Biopsy post-progression on anti-PD(L)1 (cohort A) or EGFR targeted therapy (cohort B) confirming non-squamous histology prior to study treatment initiation
* ECOG Performance Status of 0-2
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

  * ANC ≥ 1.0 x 10^9/L without granulocyte colony-stimulating factor support
  * Lymphocyte count ≥ 0.5 x 10^9/L
  * Platelet count ≥ 100 x 10^9/L without transfusion
  * Hemoglobin ≥ 80 g/L (8 g/dL) - patients may be transfused to meet this criterion.
  * AST, ALT, and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), with the following exceptions: Patients with documented liver metastases: AST and ALT ≤ 5 x ULN; Patients with documented liver or bone metastases: ALP ≤ 5 x ULN
  * Serum bilirubin ≤ 1.5 x ULN with the following exception: Patients with known Gilbert disease: serum bilirubin ≤ 3 x ULN
  * Creatinine clearance ≥ 30 mL/min (calculated using the Cockcroft-Gault formula)
  * For patients not receiving therapeutic anticoagulation: INR and aPTT ≤ 1.5 x ULN
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen defined as clinical stability on unchanged dose of therapeutic anticoagulation for ≥14 days
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 6 months after the final dose of study treatment. Women must refrain from donating eggs during this same period.
  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  * With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 6 months after the final dose of bevacizumab and 90 days after the final dose of tiragolumab. Men must refrain from donating sperm during this this same period.
  * With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of bevacizumab and 90 days after the final dose of tiragolumab to avoid potential exposure to the embryo.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of contraception.

Exclusion Criteria:

* Prior treatment with anti-TIGIT antibody therapy
* Prior treatment with anti-PD(L)1 therapeutic antibodies for advanced NSCLC (cohort B only)
* Untreated or symptomatic CNS metastases
* History of leptomeningeal disease
* Active or history of clinically significant autoimmune disease that, in the opinion of the investigator, could compromise the health and safety of the patient if treated with investigational therapy. Notable exceptions include:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen.
  * Active or history of adrenal insufficiency on stable steroid regimen.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible for the study provided all of following conditions are met: disease is well controlled at baseline and requires only low-potency topical corticosteroids; no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Known active tuberculosis
* Current treatment with anti-viral therapy for HBV
* Positive EBV viral capsid antigen antibody (IgM) testing at screening. An EBV PCR test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded.
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy other than NSCLC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death as assessed and confirmed by the study PI. Possible examples include: adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Severe infection within 3 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection (including COVID-19), bacteremia, or severe pneumonia
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the view of the investigator, contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the final dose of study treatment
* Prior immune-related adverse event resulting in permanent discontinuation of immune checkpoint blockade therapy including but not limited to anti-PD-1, anti-PD-L1 and anti-CTLA4 therapeutic antibodies (cohort A only) that, in the view of the investigator, could compromise health and safety of prospective patient if enrolled in the study
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg). Anti-hypertensive therapy to achieve these parameters is allowable
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular and cardiovascular disease (e.g., New York Heart Association Class II or greater heart failure, unstable arrhythmia, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis - including but not limited to myocardial infarction, transient ischemic attack, stroke or unstable angina) within 6 months prior to study treatment initiation
* History of hemoptysis (≥ ½ teaspoon of bright red blood per episode) or clinically significant hemorrhage within 1 month of study treatment initiation
* Evidence of bleeding diathesis or significant coagulopathy (in absence of therapeutic anticoagulation)
* Current or recent (within 10 days of first dose of study treatment) use of aspirin (>325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, < 7 days prior to the first dose of study treatment
* History of abdominal or tracheoesophageal fistula or GI perforation within 6 months prior to treatment initiation
* Clinical signs or symptoms of GI obstruction
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
* Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection. All patients with ≥ 2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection for protein
* Treatment with systemic immunosuppressive medication (including, but not limited to: corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after PI confirmation has been obtained.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 6 months after the final dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to end of treatment (average 9 months)
  As defined by investigator-assessed ORR according to RECIST v1.1

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | At the end of each cycle of therapy (every ~21 days)
  Incidence and severity of adverse events, with severity determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Progression Free Survival (PFS) | Up to 5 years
6-month PFS rate | Up to 5 years
Duration of Response (DOR) | Up to 5 years
Overall Survival (OS) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Reuss, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey